CLINICAL TRIAL: NCT06110689
Title: Capturing Physiologic Autonomic Data from Clinically Indicated Magnetic Resonance Imaging Scans in Children
Acronym: CMRI
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0400
Record Dates: First submitted 2023-10-19; First posted 2023-11-01 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Pectus Excavatum; Cardiac Anomaly
MeSH Terms: conditions — Funnel Chest; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Fontan: Patients undergoing cardiac MRI for Fontan,
  Interventions: Other: VU-AMS device
- Healthy controls: Patients undergoing thoracic MRI for chest wall deformity.
  Interventions: Other: VU-AMS device

INTERVENTIONS:
Other: VU-AMS device — Patients will wear the VU-AMS monitor prior to MRI.

SUMMARY:
The Fontan Procedure is a palliative surgical procedure used in pediatric patients with one functional ventricle. The procedure, a series of stepwise operations that alter cardiorespiratory physiology, separate the systemic and pulmonary circulations to create Fontan physiology, where the systemic venous blood flows passively and without ventricular thrust into the pulmonary circulation. The hallmark of the Fontan circulation is a sustained, abnormally elevated central venous pressure combined with decreased cardiac output, especially during periods of increased demands. Results of several studies in Fontan patients have shown reduced parasympathetic and sympathetic activity compared to controls. In children with congenital heart disease, a differential diagnosis of autonomic dysfunction may be part of their pathophysiology, a compensatory mechanism, a consequence of surgical procedures or a combination of these.

In children, measurement of ANS function is equally important. Children with single ventricle physiology (and other cardiac conditions) have routine surveillance and cardiac magnetic resonance (CMR) imaging to monitor for disease progression. While autonomic data is routinely collected and is available from these scans, these data are rarely, collected and analyzed; however, our group has shown feasibility. Therefore, autonomic data is usually unavailable in children. Despite the availability of agerelated normal values, the predictive power of autonomic activity is understudied in children and there are no published studies of quantification of autonomic data in this population.

ELIGIBILITY:
Inclusion Criteria:

* Ages 0 to ≤ 30 years
* Baseline sinus rhythm (interventricular conduction delays and bundle branch blocks allowed); and undergoing CMR scan in which sequences containing timing of aortic valve opening (cine), vector cardiogram (VCG) and respiratory bellows use will be obtained
* Fontan physiology - only for the Fontan group. Chest wall deformity or arrhythmogenic right ventricular cardiomyopathy for the healthy control group

Exclusion Criteria:

* Patient or family refusal;
* Contraindication to study procedures
* Prior participation in the study (ie, we plan to sample without replacement)

Ages: 1 Day to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients presenting for clinically indicated CMR scans with planned cine sequence and use of a respiratory bellows.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
80% availability of respiratory sinus arrhythmia from cardiac MRI (magnetic resonance imaging) | Through MRI completion up to one hour
  Data collected during MRI

OTHER OUTCOMES:
Describe difference in respiratory sinus arrhythmia in participants with Fontan | Through MRI completion up to one hour
  Collection of data from the cardiac MRI
Describe difference in respiratory sinus arrhythmia in participants with pectus | Through MRI completion up to one hour
  Collection of data from the cardiac MRI
Compare estimate of pre-ejection period (PEP) | Prior to MRI scan up to 10 minutes
  Collection of data from VU-AMS monitor
Compare estimate of pre-ejection period (PEP) | Through MRI completion up to one hour
  Collection of data from the cardiac MRI

CONTACTS AND LOCATIONS:
Overall Officials: Pornswan Ngamprasertwong, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States